CLINICAL TRIAL: NCT03440658
Title: Deficits of Strength of the Rotator Muscles of the Shoulder in Children With Sequelae of Obstetric Brachial Palsy.
Brief Title: Deficits of Strength of the Rotator Muscles of the Shoulder in Children
Acronym: ROTPOPB
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0081
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Obstetrical Brachial Plexus Palsy
Keywords: brachial plexus palsy; isokinetics; shoulder; strenght
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this retrospective work is to study the consequences of obstetrical brachial plexus paralysis on the rotator muscles of the shoulder. First of all, the investigators want to study the reproducibility of the isometric contraction forces of the rotator muscles of the shoulder thanks to an isokinetic dynamometer. The investigatorsthen want to compare the measurements obtained from the paralyzed side compared to the healthy side. The preoperative MRI performed will be studied in search of amyotrophy. These data will be compared with those of the isokinetic assessment to identify children requiring muscle transfer of reinforcement of the external rotator muscles.

DETAILED DESCRIPTION:
Obstetrical brachial plexus palsy is caused by arm stretching at birth. Recovery is not complete in a third of cases. The main sequelae is a decrease in the mobility in external rotation (ER) of the shoulder at the clinical examination. This is attributed to an imbalance between the deficient external rotator muscles (mainly infraspinatus), and the internal rotator muscles (subscapularis, pectoralis major, latissimus dorsi). A stiffness would appear because of the permanent vicious attitude of the shoulder. There is a surgical indication for arthroscopic retraction before the age of 2 years. A muscle transfer to strengthen the shoulder RE can be performed secondarily from the age of 3 years in case of persistent sequelae but the investigators lack of objective elements to ask this indication.

1. Study of the reproducibility of the isometric contraction forces of the internal and external rotator muscles obtained by isokinetic apparatus in paralyzed children.

   The isokinetic device is the gold standard for assessing muscle strength. The reproducibility of Peak Torque (PT) and Total Work (TT) will be analyzed in paralyzed children aged 3 to 5 years.
2. Comparison of isometric contraction forces of internal and external rotator muscles obtained by isokinetic device in a group of POPB children.

   Inclusion criteria: patients with obstetrical brachial plexus palsy aged between 3 and 5 years. Investigation of a significant difference in PT and TT with respect to ER and IR on the paralyzed side compared to the healthy side.
3. MRI analysis of muscular atrophy of the shoulders of paralyzed patients. The absence of recovery induces a deformation of the known shoulder joint with criteria to quantify it, but muscular amyotrophy has never been studied on the MRI of patients with brachial plexus palsy. Analysis of bilateral shoulder MRI of paralyzed patients (performed at 1 year of age as part of systematic follow-up if no-shoulder ER): describe and quantify muscle amyotrophy by measuring muscle thickness compared to healthy contralateral side. Index <0.5 in favor of amyotrophy, look for a positive correlation between the presence of muscular atrophy and joint deformity of the shoulder.
4. What are the predictive factors for recovery of external and internal shoulder rotators of children with brachial obstetrical plexus palsy?

By correlating the results of projects 1 to 3, it would be possible to:

* to identify the favorable or unfavorable prognostic factors of shoulder recovery of paralyzed children.
* identify patients with early signs of muscle recovery that do not require muscle transfer.

Perspectives: change of the therapeutic algorithm

* modification of the surgical technique according to the analysis of amyotrophy on the MRI: if subscapularis amyotrophic, more extended release with section of its upper fibers to mitigate its harmful effect on the development of the shoulder
* not to make unnecessary muscle transfer in patients with recovery of external rotator muscles masked by subscapularis fibrosis. Transfer performed if necessary secondarily according to the testing of muscular strength at the age of 3 years by isokinetic device.

ELIGIBILITY:
Inclusion criteria:

- children with obstetrical brachial plexus palsy

Exclusion criteria:

- other neurological disorders, post-traumatic shoulder stiffness

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with obstetrical brachial plexus palsy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
atrophy | 1 day
  The amyotrophy will be quantified by an index corresponding to the maximum muscle thickness measured on the MRI in T2 on the axial section passing under the spine of the scapula, between the injured side and the healthy side. This index will be measured from preoperative MRI of children. The existence of amyotrophy will be defined by an index <0.5

SECONDARY OUTCOMES:
active external or internal rotation deficit | 1 day
  active external or internal rotation deficit: measured using the iso-kinetic testing technique and defined by a maximal force moment of the injured side <70% obtained from the healthy side

CONTACTS AND LOCATIONS:
Overall Officials: Marion DELPONT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Balloufaud M, Hosni S, Bolivar J, Saguintaah M, Virassamy M, Laffont I, Coulet B, Lambert K, Delpont M. Subscapularis impairment on magnetic resonance imaging is correlated with functional limitations in neonatal brachial plexus palsy. Int Orthop. 2024 Jun;48(6):1635-1643. doi: 10.1007/s00264-023-06081-5. Epub 2024 Jan 3. PMID 38167960